CLINICAL TRIAL: NCT06277180
Title: Evaluating the Clinical Value of 68Ga-TCR-FAPI PET/CT to Guide the Surgical Treatment for Medullary Thyroid Carcinoma (MTC)
Brief Title: 68Ga-TCR-FAPI PET/CT Guided Precision Surgery for MTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCR-FAPI for MTC Surgery
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Medullary Thyroid Cancer; Prositron Emission Tomography; Fibroblast Activation Protein Inhibitor; Surgery
Keywords: Medullary Thyroid Cancer; Prositron Emission Tomography; Fibroblast Activation Protein Inhibitor; Surgery
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Newly diagnosed MTC that resect all 68Ga-TCR-FAPI-avid lesions (Experimental): Newly diagnosed MTC (did not receive previous surgery, radiotherapy or target therapy) and all pre-surgically identified 68Ga-TCR-FAPI-avid lesions are/can be successfully resected.
  Interventions: Procedure: Surgery
- Recurrent/persistent MTC that resect all 68Ga-TCR-FAPI-avid lesions (Experimental): Recurrent/persistent MTC (underwent previous surgery with currently biochemical recurrent/residual disease) and all pre-surgically identified 68Ga-TCR-FAPI-avid lesions are/can be successfully resected.
  Interventions: Procedure: Surgery
- Not all 68Ga-TCR-FAPI-avid lesions can be resected (Experimental): Not all pre-surgically identified 68Ga-TCR-FAPI-avid lesions are/can be resected.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgery is performed based on the lesion range revealed by 68Ga-TCR-FAPI PET/CT, and all 68Ga-TCR-FAPI-avid lesions are resected.
  Arms: Newly diagnosed MTC that resect all 68Ga-TCR-FAPI-avid lesions; Recurrent/persistent MTC that resect all 68Ga-TCR-FAPI-avid lesions
Procedure: Surgery — 68Ga-TCR-FAPI PET/CT identified distant metastasis or unresectable lesions, but the patient is still recommended to undergo surgery for debulking or reduce symptoms.
  Arms: Not all 68Ga-TCR-FAPI-avid lesions can be resected

SUMMARY:
This is a phase II clinical trial to evaluate the capability of 68Ga-labeled targeted covalent radiopharmaceutical (TCR) fibroblast activation protein inhibitor (FAPI) PET/CT to guide the surgical treatment of medullary thyroid carcinoma (MTC). The surgical extent of MTC is determined based on the lesion range revealed by 68Ga-TCR-FAPI PET/CT, with the main endpoint being 1-month post-surgical calcitonin level.

DETAILED DESCRIPTION:
Surgery remains the only curative option for MTC, yet the current imaging-based method (ultrasound, CT, MRI, 18F-FDG PET/CT) or calcitonin-based method are insufficient to map the extent of disease. In the previous studies, TCR-FAPI can covalently bind to FAP that increase tumor uptake and tumor retention, and better diagnosed MTC than the current radiotracers.

This is a phase II clinical trial to evaluate the capability of 68Ga-labeled targeted covalent radiopharmaceutical (TCR) fibroblast activation protein inhibitor (FAPI) PET/CT to guide the surgical treatment of medullary thyroid carcinoma (MTC). The surgical extent of MTC is determined based on the lesion range revealed by 68Ga-TCR-FAPI PET/CT, and the principles of surgery remains the same with differentiated thyroid carcinoma (i.e., lymph node dissection of level II-IV is required if lateral neck lymph node is considered metastasis). The primary endpoint of the study is 1-month post-surgical calcitonin level, and the secondary endpoints include the 2-year event free survival (EFS), the ratio of patient that change surgical plan, and the accuracy, sensitivity, specificity of 68Ga-TCR-FAPI PET/CT in identifying MTC lesions.

Patient will be divided into three arms: 1) newly diagnosed MTC and all 68Ga-TCR-FAPI PET/CT avid lesions are resected; 2) recurrent/persistent MTC and all 68Ga-TCR-FAPI PET/CT avid lesions are resected; 3) distant metastasis or unresectable lesions shown by 68Ga-TCR-FAPI PET/CT imaging but still recommended for surgical treatment. The three arms will not be compared between each other but will be separately analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years；
* Diagnosed with MTC and have surgical indication based on preliminary evaluation; the tumor may be newly diagnosed or previously treated;
* Expected survival of at least 12 weeks;
* No major organ dysfunction (heart, lung, liver, kidney and other major organ include), acute or life-threatening status of infection;
* Be willing and able to understand the research content and provide written informed consent/assent for the trial.

Exclusion Criteria:

* Have a history of imaging agent allergies;
* Does not meet the PET-CT scan sedation requirements, or has contraindications for PET-CT examination;
* Be pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial;
* No surgical indication (i.e., no measurable disease, unresectable disease, or significant present of distant metastasis), refusing surgery or 68Ga-TCR-FAPI PET/CT-guided surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-month post-surgery calcitonin level | 1-month post-surgery
  1-month post-surgery calcitonin level

SECONDARY OUTCOMES:
2-year event free survival | 2-year post-surgery
  2-year event free survival
Ratio of patient that change surgical plan | immediately after surgery
  Ratio of patient that change surgical plan
Accuracy, sensitivity, specificity of 68Ga-TCR-FAPI PET/CT in identifying MTC lesions | 1-month post-surgery
  Accuracy, sensitivity, specificity of 68Ga-TCR-FAPI PET/CT in identifying MTC lesions

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No